CLINICAL TRIAL: NCT04496804
Title: BIPAMS-Brain:Examining the Neural Effects of a Behavioral Intervention for Physical Activity in Multiple Sclerosis
Brief Title: Examining the Neural Effects of a Behavioral Intervention for Physical Activity in Multiple Sclerosis
Acronym: BIPAMS-Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert W Motl, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 300005111
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: physical activity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Behavior Therapy; Exercise; Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention for Physical Activity in MS (BIPAMS) (Experimental): The current behavioral intervention consists of two primary components; an Internet website and one-on-one video chats with a behavioral coach. The Internet website involves content delivered through interactive video courses. The interactive video courses are based on elements of social cognitive theory. Each courses consists of an introduction, the primary content, and a take home message. The interactive courses include embedded, supplementary options such as videos on content and worksheets related to the topic. A pedometer is provided for tracking steps, and these steps will be entered into the website so progress can be monitored. The chats support adherence to the intervention, discussion of website material, supportive accountability, and reporting of adverse events/injuries. The chats are conducted face-to-face through Skype. The chats occur 7 times during the first 2 months, 4 times during the second 2 months, and twice during the final 2 months of the intervention.
  Interventions: Behavioral: Behavioral Intervention for Physical Activity in MS (BIPAMS)
- Wellness for MS (WellMS) (Sham Comparator): Provides an Internet website and one-on-one video chats that discuss materials about self-managing multiple sclerosis (MS) consequences and health indicators through methods other than physical activity. The materials are transformations of brochures provided by the National MS Society, including Gait or Walking Problems: The Basic Facts; MS and Your Emotions; Pain: The Basic Facts; Solving Cognitive Problems; Taming Stress in MS; Food for Thought: MS and Nutrition; and Vitamins, Minerals, and Herbs: An Introduction. The delivery of the Internet materials and chat sessions will occur on the same time schedule and frequency as the intervention condition, and will have a comparable time commitment. The control condition will not involve tracking steps and a pedometer with not be provided.
  Interventions: Behavioral: Wellness for MS (WellMS)

INTERVENTIONS:
Behavioral: Behavioral Intervention for Physical Activity in MS (BIPAMS) — A behavioral intervention that involves an Internet website and one-on-one video coaching calls for increasing physical activity in people with MS.
  Arms: Behavioral Intervention for Physical Activity in MS (BIPAMS)
Behavioral: Wellness for MS (WellMS) — A behavioral intervention that involves an Internet website and one-on-one video coaching calls for increasing wellness in people with MS.
  Arms: Wellness for MS (WellMS)

SUMMARY:
Multiple sclerosis [MS] is a prevalent neurological disease that is the leading cause of irreversible neurological disability among young women and the second leading cause of disability among young men in the United States. This disease results in the progressive loss of walking mobility and substantial worsening of cognition, symptoms, and quality of life over time. There is evidence that physical activity is beneficially associated with aerobic fitness and brain structure and function in persons with MS. Nevertheless, this population is strikingly sedentary and physically inactive. This highlights a vital opportunity to improve aerobic fitness and brain health by developing behavioral interventions that increase physical activity. To that end, this project is a Phase-II randomized control trial for examining the efficacy of a behavioral intervention that is based on social-cognitive theory and delivered through the Internet for increasing physical activity and, secondarily, improving aerobic fitness and brain structure and function in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis
* relapse free in the last 30 days
* being non-active defined as not engaging in regular activity (30 minutes accumulated per day) on more than 2 days of the week during the previous 6 months
* ambulate without assistance
* low risk for contraindications for MRI

Exclusion Criteria:

* moderate or high risk for undertaking strenuous or maximal exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate to vigorous physical activity - Baseline | Assessment will be conducted before the intervention
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.
Minutes of moderate to vigorous physical activity - Post intervention | Assessment will be conducted immediately after the intervention
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.

SECONDARY OUTCOMES:
cardiorespiratory fitness; oxygen consumption during exercise - baseline | Assessment will be conducted before the intervention
  A graded exercise test on a treadmill. Participants will walk at a quick pace on the treadmill and the incline will increase every 2 minutes until the participant is no longer able to keep pace with the treadmill.
cardiorespiratory fitness; oxygen consumption during exercise - post intervention | Assessment will be conducted immediately after the intervention
  A graded exercise test on a treadmill. Participants will walk at a quick pace on the treadmill and the incline will increase every 2 minutes until the participant is no longer able to keep pace with the treadmill.
distance walked - baseline | Assessment will be conducted before the intervention
  The six-minute walk test will be used to measure walking endurance. The test involves walking for 6 minutes without stopping.
distance walked - post-intervention | Assessment will be conducted immediately after the intervention
  The six-minute walk test will be used to measure walking endurance. The test involves walking for 6 minutes without stopping.
information processing speed; cognitive function - baseline | Assessment will be conducted before the intervention
  The symbol digit modalities test will be used to measure information processing speed. The test involves matching numbers to symbols.
information processing speed; cognitive function - post intervention | Assessment will be conducted immediately after the intervention
  The symbol digit modalities test will be used to measure information processing speed. The test involves matching numbers to symbols.
volume of subcortical grey matter brain structures - baseline | Assessment will be conducted before the intervention
  An MRI will be conducted to measure brain structure.
volume of subcortical grey matter brain structures - post intervention | Assessment will be conducted immediately after the intervention
  An MRI will be conducted to measure brain structure.
resting state functional brain connectivity - baseline | Assessment will be conducted before the intervention
  An MRI will be conducted to measure brain function.
resting state functional brain connectivity - post intervention | Assessment will be conducted immediately after the intervention
  An MRI will be conducted to measure brain function.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Motl, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States